CLINICAL TRIAL: NCT06043453
Title: Revitalization of Immature Permanent Teeth With or Without Apical Periodontitis Post Trauma: a European Multicenter Cohort Study
Brief Title: Revitalization of Traumatized Immature Permanent Teeth
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: University Ghent (Other); University of Erlangen-Nürnberg (Other); University of Regensburg (Other); University of Coimbra (Other)
Responsible Party: Sponsor
Other Study IDs: S67181
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2023-08

CONDITIONS: Apical Periodontitis; Trauma
MeSH Terms: conditions — Periapical Periodontitis; Wounds and Injuries | interventions — Air Conditioning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with AP
  Interventions: Other: revitalization
- without AP
  Interventions: Other: revitalization

INTERVENTIONS:
Other: revitalization — The main idea behind revitalization is to firstly disinfect the root canal and subsequently attract or transplant mesenchymal stem cells from the (remaining) dental pulp and apical papilla (in case of immature permanent teeth) into the root canal. More specifically, this therapy is not based on mechanical and (aggressive) chemical debridement as in conventional root canal treatment but is supported by the pillars of tissue engineering: stem cells, growth factors and a scaffold .

SUMMARY:
This study aims to assess the hypothesis that revitalization of teeth without (a)symptomatic apical periodontitis have a more favourable outcome in terms of further root development, periapical bone healing, maintaining/regaining pulp sensitivity and survival, than teeth with (a)symptomatic apical periodontitis.

DETAILED DESCRIPTION:
1. Trial objectives

   This study aims to investigate the effectiveness of revitalization procedures, in terms of maintaining or restoring periapical health, further root development and regaining of pulp sensitivity, in immature permanent teeth with (group 1) or without (group 2) (a)symptomatic apical periodontitis .
2. Primary endpoints RRA at 1 year post revitalization. 3 Secondary endpoints Maintained or restored periapical health (evaluated within each group separately due to expected baseline inequivalency between groups) 1 year post revitalization.

4 Other endpoints

* RRA 2 and 3 years post revitalization
* Maintained or restored periapical health 2 and 3 years post revitalization (evaluated within each group separately)
* Pulp sensitivity 1-3 years post revitalization (evaluated within each group separately due to expected baseline inequivalency between groups)
* Tooth survival 3 years post revitalization (even if no further root development and incomplete periapical bone healing with no clinical symptoms).

  5 Trial Design Open, prospective cohort, multicenter Blinded: radiographic assessment and statistical analysis; operators and patients cannot be blinded, due to practically not feasible.

ELIGIBILITY:
Inclusion Criteria:

* Provision of Informed Consent
* Female and male patients
* Age range: 6-18 years
* "Healthy": ASA I and II
* Permanent immature tooth (Cvek stage of root maturation ≤ 2) requiring revitalization
* Etiological factor: (a)symptomatic apical periodontitis post dental trauma or irreversible pulpitis post dental trauma

Exclusion Criteria:

* Unlikely to be able to comply with the study procedures, as judged by the investigator
* Patients older than 18 years and younger than 6
* Deciduous teeth
* Cvek root maturation stage > 2: permanent immature tooth that can be treated by conventional root canal treatment or apexification
* Known or suspected current malignancy
* History of chemotherapy within 5 years prior to study
* History of radiation in the head and neck region
* History of other metabolic bone diseases
* Bleeding disorders
* Involvement in the planning and conduct of the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy patients (ASA I and II), younger than 18 years, presenting an immature permanent tooth in need of treatment, etiological factor: (a)symptomatic apical periodontitis or irreversible pulpitis post dental trauma, no other endodontic treatment option than revitalization possible.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
radiographic root area (RRA) | 1 year
  RRA post revitalization

SECONDARY OUTCOMES:
periapical health | 1 year
  Maintained or restored periapical health post revitalization

OTHER OUTCOMES:
RRA 2 and 3 years post revitalization | 2 and 3 years
  RRA post revitalization
Maintained or restored periapical health 2 and 3 years post revitalization (evaluated within each group separately) | 2 and 3 years
  periapical health
Pulp sensitivity 1-3 years post revitalization (evaluated within each group separately due to expected baseline inequivalency between groups) | 1 to 3 years
  pulp sensitivity
Tooth survival 3 years post revitalization (even if no further root development and incomplete periapical bone healing with no clinical symptoms). | 3 years
  tooth survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No